CLINICAL TRIAL: NCT03801876
Title: Phase III Randomized Trial of Proton Beam Therapy (PBT) Versus Intensity Modulated Photon Radiotherapy (IMRT) for the Treatment of Esophageal Cancer
Brief Title: Comparing Proton Therapy to Photon Radiation Therapy for Esophageal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI006; NCI-2018-03378 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GI006 (Other: NRG Oncology); NRG-GI006 (Other: CTEP); U10CA180822 (NIH); U10CA180868 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage I Esophageal Adenocarcinoma AJCC v8; Clinical Stage I Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage I Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Thoracic Esophagus Squamous Cell Carcinoma
MeSH Terms: interventions — Specimen Handling; Capecitabine; Carboplatin; Docetaxel; Esophagectomy; Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated; Leucovorin; Oxaliplatin; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (PBT, concurrent chemotherapy, esophagectomy) (Experimental): Patients undergo PBT over 28 fractions 5 days a week for 5.5 weeks. Patients also receive chemotherapy consisting of carboplatin/paclitaxel, or FOLFOX/CAPOX, or docetaxel/5-FU (with capecitabine an acceptable substitute for 5-FU) as determined by the patient and their treating physician while undergoing PBT. Additionally, patients undergo blood sample collection, and PET/CT or CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Capecitabine; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Esophagectomy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (IMRT, concurrent chemotherapy, esophagectomy) (Active Comparator): Patients undergo IMRT over 28 fractions 5 days a week for 5.5 weeks. Patients also receive chemotherapy consisting of carboplatin/paclitaxel, or FOLFOX/CAPOX, or docetaxel/5-FU (with capecitabine an acceptable substitute for 5-FU) as determined by the patient and their treating physician while undergoing IMRT. Additionally, patients undergo blood sample collection, and PET/CT or CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Capecitabine; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Esophagectomy; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Oral
  Other Names: Ro 09-1978/000; Xeloda
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Docetaxel — IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Procedure: Esophagectomy — Undergo esophagectomy
  Other Names: excision of the esophagus
Drug: Fluorouracil — IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Group II (IMRT, concurrent chemotherapy, esophagectomy)
Drug: Leucovorin Calcium — Oral
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Proton Beam Radiation Therapy — Undergo PBT
  Other Names: External beam radiation therapy protons (procedure); External Beam Radiotherapy (protons); PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; PROTON Therapy; Radiation, Proton Beam
  Arms: Group I (PBT, concurrent chemotherapy, esophagectomy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well proton beam radiation therapy compared with intensity modulated photon radiotherapy works in treating patients with stage I-IVA esophageal cancer. Proton beam radiation therapy uses a beam of protons (rather than x-rays) to send radiation inside the body to the tumor without damaging much of the healthy tissue around it. Intensity modulated photon radiotherapy uses high-energy x-rays to deliver radiation directly to the tumor without damaging much of the healthy tissue around it. It is not yet known whether proton beam therapy or intensity modulated photon radiotherapy will work better in treating patients with esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if overall survival (OS) is improved with proton beam radiation therapy (PBT) treatment as compared to intensity modulated photon radiation therapy (IMRT) as part of planned protocol treatment for patients with esophageal cancer.

II. To determine if OS with PBT is non-inferior to IMRT as part of planned protocol treatment and that there will be less grade 3+ cardiopulmonary toxicity with PBT than with IMRT.

SECONDARY OBJECTIVES:

I. To compare the symptom burden and impact on functioning of patients between treatment modalities based on Patient Reported Outcome (PRO) measures of symptoms using MD Anderson Symptom Inventory (MDASI) and Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue.

II. To compare the Quality-Adjusted Life Years (QALY) using EuroQol five-dimensional questionnaire (EQ5D) as a health outcome between PBT and IMRT, if the protocol primary endpoint is met.

III. To assess the pathologic response rate between PBT and IMRT. IV. To assess the cost-benefit economic analysis of treatment between radiation modalities.

V. To compare the length of hospitalization after protocol surgery between PBT and IMRT.

VI. To compare the incidence of grade 4 lymphopenia during chemoradiation between PBT and IMRT.

VII. To compare lymphocyte nadir at first follow-up visit after completion of chemoradiation between PBT & IMRT.

VIII. To estimate the locoregional failure, distant metastatic free survival, and progression-free survival of patients treated with PBT versus IMRT.

IX. To compare incidence of both early (< 90 days from treatment start) and late (≥ 90 days from treatment start) cardiovascular and pulmonary events between PBT versus IMRT.

X. To compare the total toxicity burden (TTB) of IMRT versus PBT based on a composite index of 9 individual cardiopulmonary toxicities.

EXPLORATORY OBJECTIVES:

I. To collect biospecimens for future analyses, for example to assess cardiac and inflammatory biomarkers in association with treatment complications.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo PBT over 28 fractions 5 days a week for 5.5 weeks. Patients also receive chemotherapy consisting of carboplatin/paclitaxel, or fluorouracil/leucovorin calcium/oxaliplatin (FOLFOX)/capecitabine-oxaliplatin (CAPOX), or docetaxel/fluorouracil (5-FU, with capecitabine an acceptable substitute for 5-FU), as determined by the patient and their treating physician while undergoing PBT.

GROUP II: Patients undergo IMRT over 28 fractions 5 days a week for 5.5 weeks. Patients also receive chemotherapy consisting of carboplatin/paclitaxel, or FOLFOX/CAPOX, or docetaxel/5-FU (with capecitabine an acceptable substitute for 5-FU) as determined by the patient and their treating physician while undergoing IMRT.

In both groups, within 4-8 weeks after completion of chemotherapy and radiation therapy, patients should undergo an esophagectomy if it's determined that the patient can tolerate an esophagectomy and whether the tumor is surgically resectable.

Additionally, patients undergo blood sample collection, and positron emission tomography (PET)/computed tomography (CT) or CT throughout the study.

After completion of study treatment, patients are followed up every 3-6 months for 3 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* Histologically proven diagnosis of adenocarcinoma or squamous cell carcinoma of the thoracic esophagus or gastroesophageal junction (Siewert I-II)
* Stage I-IVA, excluding T4b, according to the American Joint Committee on Cancer (AJCC) 8th edition based on the following diagnostic workup:

  * History/physical examination
  * Whole-body fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) with or without contrast (preferred) or chest/abdominal (include pelvic if clinically indicated) CT with contrast

    * For patients who DID NOT receive induction chemotherapy, scan must occur within 30 days prior to Step 1 registration
    * For patients who DID receive induction chemotherapy, scan must occur:

      * Within 30 days after final induction chemotherapy dose; OR
      * Within 30 days prior to Step 1 registration
    * Note: Patients who had prior endoscopic mucosal resection (EMR) with a diagnosis of AJCC stage I-IVA, excluding T4b, esophageal cancer are eligible
* Surgical consultation to determine whether or not the patient is a candidate for resection after completion of chemoradiation
* Induction chemotherapy for the current malignancy prior to concurrent chemoradiation allowed if last dose is no more than 90 days and no less than 10 days prior to Step 1 registration; only FOLFOX, CAPOX, durvalumab-fluorouracil, leucovorin, oxaliplatin and docetaxel (FLOT) (D-FLOT) and FLOT will be allowed as the induction chemotherapy regimen
* Age ≥ 18
* Zubrod performance status 0, 1, or 2
* Absolute neutrophil count (ANC) (within 30 days prior to Step 1 registration)

  * For patients who DID NOT receive induction chemotherapy: ANC ≥ 1,500 cells/mm^3
  * For patients who DID receive induction chemotherapy: ANC ≥ 1,000 cells/mm^3
* Platelets (within 30 days prior to Step 1 registration)

  * For patients who DID NOT receive induction chemotherapy: Platelets ≥ 100,000/uL
  * For patients who DID receive induction chemotherapy: Platelets ≥ 75,000/uL
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable) (within 30 days prior to Step 1 registration)
* Serum creatinine ≤ 1.5 X upper limit of normal (ULN) or creatinine clearance > 40 mL/min estimated by Cockcroft-Gault formula (within 30 days prior to Step 1 registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (within 30 days prior to Step 1 registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN (within 30 days prior to Step 1 registration)
* Negative pregnancy test (serum or urine) within 14 days prior to Step 1 registration for women of child bearing potential
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Cervical esophageal cancers arisen from 15-18 cm from the incisors
* Patients with T4b disease according to the AJCC 8th edition
* Definitive clinical or radiologic evidence of metastatic disease
* Any active malignancy within 2 years of study registration that may alter the course of esophageal cancer treatment
* Prior thoracic radiotherapy that would result in overlap of radiation therapy fields
* Severe, active co-morbidity defined as follows:

  * Active uncontrolled infection requiring IV antibiotics at the time of Step 1 registration
  * Uncontrolled symptomatic congestive heart failure, unstable angina, or cardiac arrhythmia not controlled by any device or medication at the time of Step 1 registration
  * Myocardial infarction within 3 months prior to Step 1 registration
* Pregnant and/or nursing females
* Human immunodeficiency virus (HIV) positive with CD4 count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 30 days prior to registration. Note also that HIV testing is not required for eligibility for this protocol. This exclusion criterion is necessary because the treatments involved in this protocol may be significantly immunosuppressive
* PRIOR TO STEP 2 REGISTRATION:
* Unable to obtain confirmation of payment coverage (insurance or other) for either possible radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2031-12-21 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death due to any cause or date of last follow-up for patients without an OS event reported. This analysis occurs after 173 deaths; estimated to occur 4 years after accrual completion
  Will be estimated by the Kaplan-Meier method. The distributions of OS between treatment arms will be compared using the log rank test.
Incidence of specific grade 3+ cardiopulmonary adverse events (AEs) that are definitely, probably, or possibly related to protocol treatment | From baseline up to 8 years
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Difference in proportion of defined cardiopulmonary AEs will be analyzed with a chi-squared test.

SECONDARY OUTCOMES:
Change in patient reported outcomes (PROs) of symptom and function | Baseline up to 12 months after end of chemoradiation
  Will be assessed using the MD Anderson Symptom Inventory (MDASI) and the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue tools. The primary analysis cohorts for PRO endpoints will be intent-to-treat, with sensitivity analyses done limited to patients that started protocol treatment. General linear models with maximum likelihood estimation will be used to assess MDASI symptom severity and functioning trends across time as the primary PRO endpoints. Mean change (follow-up time point - baseline score) in fatigue will be compared between treatment arms using a t-test. If the data do not satisfy the normality assumption, a Wilcoxin test may be used instead. Additionally, a general linear model with maximum likelihood estimation will be used to assess fatigue trends across time.
Pathologic response rate | At time of surgery
  A Chi-square test will be used to compare the pathologic response rates between the treatment arms.
Length of hospitalization | From baseline up to 8 years
  Will be defined as number of days in the hospital post protocol-defined surgery. Mean hospitalization days will be compared between treatment arms using a t-test. If the data do not satisfy the normality assumption, a Wilcoxin test may be used instead.
Grade 4 lymphopenia during chemoradiation | From baseline up to 8 years
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients experiencing grade 4 lymphopenia during chemoradiation will be compared between treatment arms using a chi-squared test.
Lymphocyte counts | From baseline up to 8 years
  Mean lymphocyte counts at first post chemoradiation follow-up will be compared between treatment arms using a t-test. If the data do not satisfy the normality assumption, a Wilcoxin test may be used instead.
Locoregional failure (LRF) | From the date of randomization to the date of first LRF or date of last follow-up for patients without an LRF event reported, assessed up to 8 years
  Will be defined as local/regional recurrence or progression. Will be estimated by the cumulative incidence method, with death as a competing risk. The distribution of LRF estimates between the two arms will be compared using Gray's test. The Fine-Gray regression model will be used to analyze the effects of factors, in addition to treatment, which may be associated with LRF.
Distant metastatic-free survival (DMFS) | From the date of randomization to the date of first DMFS failure or last follow-up for patients without a reported DMFS event, assessed up to 8 years
  Will be defined as appearance of distant metastasis or death due to any cause. Will be estimated by the Kaplan-Meier method and estimates between the two treatment arms will be compared using the log rank test. The Cox proportional hazard regression model will be used to analyze the effects of factors, in addition to treatment, which may be associated with DMFS.
Progression-free survival | From the date of randomization to the date of first PFS failure or last follow-up for patients without a reported PFS event, assessed up to 8 years
  Will be defined as appearance of local/regional/distant failure or death due to any cause. Will be estimated by the Kaplan-Meier method and estimates between the two treatment arms will be compared using the log rank test. The Cox proportional hazard regression model will be used to analyze the effects of factors, in addition to treatment, which may be associated with PFS.
Quality-adjusted life years (QALY) | Assessed up to 8 years
  Will be evaluated and compared using EuroQol five-dimensional questionnaire (EQ-5D) only if the primary endpoint is met.
Cost-benefit economic analysis of treatment | Assessed up to 8 years
  Will be calculated by the visual analog scale (VAS) and index scores form the EQ-5D-5L only be done if primary endpoint is met. Will be compared between treatment arms using a t-test with a 2-sided significance level of 0.05. If there are significant differences, then a cost analysis will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Lin, Principal Investigator — NRG Oncology
Locations (95):
- United States (95):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Alton Memorial Hospital, Alton, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Radiation Therapy-Northfield, Northfield, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - New York Proton Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thompson Proton Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Thompson Oncology Group-Maryville, Maryville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin